CLINICAL TRIAL: NCT01617668
Title: A Phase II Multi-center, Open-label, Neoadjuvant, Randomized Study of Weekly Paclitaxel With or Without LCL161 in Patients With Triple Negative Breast Cancer
Brief Title: A Randomized, Phase 2, Neoadjuvant Study of Weekly Paclitaxel With or Without LCL161 in Patients With Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLCL161A2201; 2012-000677-23 (EudraCT Number)
Record Dates: First submitted 2012-05-30; First posted 2012-06-12 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer,; LCL161,; paclitaxel,; neoadjuvant,; triple negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — LCL161; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel with LCL161 (Experimental): Patients randomized to the experimental arm received paclitaxel 80 mg/m2 weekly + LECL161 1800 mg once weekly for 12 weeks. Equal numbers of patients with gene expression signature positive and negative disease were included in each treatment arm.
  Interventions: Drug: LCL161; Drug: paclitaxel
- Paclitaxel without LCL161 (Active Comparator): Patients randomized to the control arm received paclitaxel 80 mg/m2 weekly for 12 weeks. Equal numbers of patients with gene expression signature positive and negative disease were included in each treatment arm.
  Interventions: Drug: paclitaxel

INTERVENTIONS:
Drug: LCL161 — LCL161 was available as 300 mg, tablets, which was supplied in child-resistant bottles.
  Arms: Paclitaxel with LCL161
Drug: paclitaxel — Commercially available paclitaxel was sourced locally by each study site. Generic paclitaxel could be used for study treatment.
  iv 80mg/m2

SUMMARY:
To assess whether adding LCL161 to weekly paclitaxel enhances the efficacy of paclitaxel in women with triple negative breast cancer whose tumors are positive for a defined pattern of gene expression

DETAILED DESCRIPTION:
This is a phase 2, randomized, two-arm, open-label, neoadjuvant, multicenter study in newly diagnosed women with triple-negative breast cancer. Eligible patients will be limited to those with clinical stages T2, N0-N2, M0.

For those patients with triple-negative disease identified on diagnostic biopsy, the presence or absence of the gene expression signature will be determined in a molecular pre-screening phase using the diagnostic biopsy material; patients with TNBC that are positive and negative for the gene expression signature will be eligible for enrollment.

Following a Screening/baseline period to determine eligibility, patients will be randomized to either paclitaxel 80 mg/m2 IV given weekly (the control arm) or paclitaxel 80 mg/m2 IV weekly immediately followed by LCL161 1800 mg PO once weekly (the experimental arm). Enrollment on these arms will be balanced within regions of the world and are stratified 1:1 for gene expression signature status. Treatment will be administered each week for 12 weeks (4 cycles). The length of each treatment cycle is 21 days.

A total of 200 patients will be enrolled and treated, 100 patients in each treatment arm of the study; each arm will contain 50 patients with gene expression signature positive disease and 50 patients with gene expression signature negative disease.

An interim analysis is planned for this study when approximately 50 patients with gene expression signature positive disease have been treated and have either completed the study and have undergone surgery, or have permanently discontinued study treatment for any reason.

For all patients, a tumor biopsy will be performed approximately 24 hours after the first or second dose of study treatment (paclitaxel or paclitaxel + LCL161) to compare the extent of apoptosis in tumor treated with control or experimental therapy. Patients will be scheduled for breast-conserving surgery or mastectomy 15 weeks plus a window of not more than 1 week from the date the subject receives her first treatment (no more than 16 weeks after first treatment). All treated patients are planned to undergo surgery. However, to evaluate the presence of persistent disease those patients with apparent substantial residual or progressive disease or who do not undergo surgery for any reason must have a core needle biopsy of the primary tumor after completing study treatment. At the completion of study treatment, patients are expected to continue post-operative treatment with a standard anthracycline-based chemotherapy regimen such as FAC (5-FU/doxorubicin/cyclophosphamide), FEC (5-FU/epirubicin/cyclophosphamide) or AC (doxorubicin/cyclophosphamide). The specific regimen will be chosen by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of invasive triple negative breast cancer
* Known status for the LCL161 predictive gene expression signature as determined during molecular pre-screening
* Candidates for mastectomy or breast-conserving surgery
* Primary tumor of greater than 20 mm and less than or equal to 50 mm diameter measured by imaging (previous Amendment #3 was tumor size greater than 10 mm)
* Regional nodes N0-N2
* Absence of distant metastatic disease
* ECOG performance status 0-1
* Adequate bone marrow function
* Adequate liver function and serum transaminases
* Adequate renal function

Exclusion Criteria:

* Bilateral or inflammatory breast cancer (bilateral mammography is required during Screening/baseline); locally recurrent breast cancer
* Patients currently receiving systemic therapy for any other malignancy, or having received systemic therapy for a malignancy in the preceding 3 months
* Uncontrolled cardiac disease
* Patients who are currently receiving chronic treatment (>3 months) with corticosteroids at a dose ≥ 10 mg of prednisone (or its glucocorticoid equivalent) per day (inhaled and topical steroids are allowed), or any other chronic immunosuppressive treatment that cannot be discontinued prior to starting study drug
* Impaired GI function that may affect the absorption of LCL161
* Pregnant or breast feeding (lactating) women
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 180 days after study treatment
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2012-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (45):
- United States (13):
  - Highlands Oncology Group Dept of Highlands Oncology Grp, Fayetteville, Arkansas
  - Cedars Sinai Medical Center SC, Los Angeles, California
  - University of California at Los Angeles UCLA SC, Los Angeles, California
  - Stanford University Medical Center Stanford, Stanford, California
  - Yale University School of Medicine Yale Univ, New Haven, Connecticut
  - H. Lee Moffitt Cancer Center & Research Institute H. Lee Moffitt SC, Tampa, Florida
  - Massachusetts General Hospital Mass General 2, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center Dept Onc, New York, New York
  - Ohio State Comprehensive Cancer Center/James Cancer Hospital Ohio State, Columbus, Ohio
  - Vanderbilt University Medical Center Vanderbilt - Thompson Ln, Nashville, Tennessee
  - Baylor College of Medicine Dept of Oncology, Houston, Texas
  - Cancer Therapy & Research Center / UT Health Science Center InstituteForDrugDevelopment(5), San Antonio, Texas
  - University of Wisconsin / Paul P. Carbone Comp Cancer Center Univ Wisc 2, Madison, Wisconsin
- Novartis Investigative Site, Nedlands, Western Australia, Australia
- Brazil (2):
  - Novartis Investigative Site, Itajaí, Santa Catarina
  - Novartis Investigative Site, São Paulo, São Paulo
- Czechia (2):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Olomouc
- Germany (10):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, München
- Ireland (2):
  - Novartis Investigative Site, Dublin, Ireland
  - Novartis Investigative Site, Dublin
- Novartis Investigative Site, Padua, PD, Italy
- Novartis Investigative Site, Saint Petersburg, Russia
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (5):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Valencia, Valencia
- Taiwan (3):
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Kuei-Shan Chiang, Taoyuan/ Taiwan ROC
- United Kingdom (4):
  - Novartis Investigative Site, Brighton, East Sussex
  - Novartis Investigative Site, Kingston upon Thames, Surrey
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 215 patients were randomized to receive the study treatment. 105 gene expression signature positive patients were randomized to LCL161+paclitaxel (N=51) or paclitaxel only (N=54). 110 gene expression signature negative patients were randomized to LCL161+paclitaxel (N=55) or paclitaxel only (N=55).
Pre-assignment Details: Only 50 of 54 pts in the Paclitaxel without LCL161 (Positive group) received study drug; Only 53 of 55 pts in the Paclitaxel without LCL161 (Negative group) received study drug.
Groups:
- Paclitaxel With LCL161 (Positive Group): Patients randomized to the experimental arm received paclitaxel 80 mg/m2 weekly + LECL161 1800 mg once weekly for 12 weeks. Equal numbers of patients with gene expression signature positive and negative disease were included in each treatment arm.
- Paclitaxel Without LCL161 (Positive Group); Paclitaxel Without LCL161 (Negative Group): Patients randomized to the control arm received paclitaxel 80 mg/m2 weekly for 12 weeks. Equal numbers of patients with gene expression signature positive and negative disease were included in each treatment arm.
- Paclitaxel With LCL161 (Negative Group): Patients randomized to the experimental arm received paclitaxel 80 mg/m2 weekly + LCL161 1800 mg once weekly for 12 weeks. Equal numbers of patients with gene expression signature positive and negative disease were included in each treatment arm.
Period: Overall Study
Arm/Group | Paclitaxel With LCL161 (Positive Group) | Paclitaxel Without LCL161 (Positive Group) | Paclitaxel With LCL161 (Negative Group) | Paclitaxel Without LCL161 (Negative Group)
Started | 51 | 50 (54 patients were randomized and only 50 received study treatment.) | 55 | 53 (55 patients were randomized and only 53 received study treatment.)
Randomized Patients | 51 | 54 | 55 | 55
Completed | 38 | 41 | 32 | 38
Not Completed | 13 | 9 | 23 | 15
Not completed — Adverse Event | 7 | 0 | 12 | 5
Not completed — Physician Decision | 1 | 2 | 3 | 0
Not completed — Progressive Disease | 4 | 4 | 6 | 9
Not completed — Subject/guardian decision | 1 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) was composed of all patients who received at least one full or partial dose of LCL161 + paclitaxel or one full or partial dose of paclitaxel alone.
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel With LCL161 | Paclitaxel Without LCL161 | Total
Number analyzed (Participants) | 106 | 103 | 209
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.6 (10.14) | 48.7 (9.98) | 48.7 (10.04)
Age, Customized [Number; unit: Participants]
  < 65 years | 98 | 96 | 194
  >= 65 years | 8 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 103 | 209
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR) Rate in Breast After 12 Weeks of Therapy
Description: pCR rate was defined as histopathologically confirmed absence of invasive disease in the breast. To assess whether adding LCL161 to weekly paclitaxel enhances the efficacy of paclitaxel in women with triple negative breast cancer. Analyses were performed separately in the gene expression signature negative and positive groups. This analysis was based on Bayesian design using a binomial distribution for the data with a beta prior. The measurement type used for this analysis is posterior median and the method of dispersion is Credible Interval (Crl) and not Confidence Interval (CI). Median values are posterior medians of pCR rate for each group.
Time Frame: 12 weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Percentage of Participants
Groups:
- LCL161 + Paclitaxel (Gene Expression Signature Positive): Patients randomized to the experimental arm for gene expression signature positive received LCL161 1800 mg once weekly + paclitaxel 80 mg/m2 weekly for 12 weeks. Equal numbers of patients with gene expression signature positive and negative disease were included in each treatment arm.
- Paclitaxel Only (Gene Expression Signature Positive): Patients randomized to the control arm for gene expression signature positive received paclitaxel 80 mg/m2 weekly for 12 weeks. Equal numbers of patients with gene expression signature positive and negative disease were included in each treatment arm.
- LCL161 + Paclitaxel (Gene Expression Signature Negative): Patients randomized to the experimental arm for gene expression signature negative received paclitaxel 80 mg/m2 weekly + LCL161 1800 mg once weekly for 12 weeks. Equal numbers of patients with gene expression signature positive and negative disease were included in each treatment arm.
- Paclitaxel Only (Gene Expression Signature Negative): Patients randomized to the control arm for gene expression signature negative received paclitaxel 80 mg/m2 weekly for 12 weeks. Equal numbers of patients with gene expression signature positive and negative disease were included in each treatment arm.
Arm/Group | LCL161 + Paclitaxel (Gene Expression Signature Positive) | Paclitaxel Only (Gene Expression Signature Positive) | LCL161 + Paclitaxel (Gene Expression Signature Negative) | Paclitaxel Only (Gene Expression Signature Negative)
Number analyzed (Participants) | 51 | 50 | 55 | 53
Percentage of Participants | 24.9 [14.5 to 37.8] | 23.4 [13.3 to 36.2] | 6.9 [2.2 to 15.5] | 9.1 [3.3 to 18.6]

2. Primary Outcome: Number of Participants With Pathological Complete Response (pCR) in Breast After 12 Weeks of Therapy
Description: To assess the number of patients who experienced a pathological response in breast.
Time Frame: 12 weeks
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | LCL161 + Paclitaxel (Gene Expression Signature Positive) | Paclitaxel Only (Gene Expression Signature Positive) | LCL161 + Paclitaxel (Gene Expression Signature Negative) | Paclitaxel Only (Gene Expression Signature Negative)
Number analyzed (Participants) | 51 | 50 | 55 | 53
Participants | 13 [14.5 to 37.8] | 12 [13.3 to 36.2] | 4 [2.2 to 15.5] | 5 [3.3 to 18.6]

3. Primary Outcome: Difference in pCR Rates Between Treatment Arms
Description: pCR rate was defined as histopathologically confirmed absence of invasive disease in the breast. To assess whether adding LCL161 to weekly paclitaxel enhances the efficacy of paclitaxel in women with triple negative breast cancer. Analyses were performed separately in the gene expression signature negative and positive groups. This analysis was based on the posterior distribution of the difference in pCR rates between the experimental and control arms of the study, within each gene expression signature group.The measurement type used for this analysis is posterior median and the method of dispersion is Credible Interval (Crl) and not Confidence Interval (CI). 95% Confidence interval is actually 95% credible interval.
Time Frame: 12 weeks
Population: FAS are patients who received at least 1 full or partial dose of LCL161 + paclitaxel or 1 full or partial dose of paclitaxel alone. These values are medians of posterior distribution of difference of pCR rate between treatment arms based on a Bayesian model. 95% Confidence interval is actually 95% credible interval.
Measure: Median (95% Confidence Interval); unit: Difference in percentage of participants
Arm/Group | LCL161 + Paclitaxel (Gene Expression Signature Positive) | Paclitaxel Only (Gene Expression Signature Positive) | LCL161 + Paclitaxel (Gene Expression Signature Negative) | Paclitaxel Only (Gene Expression Signature Negative)
Number analyzed (Participants) | 51 | 50 | 55 | 53
Difference in percentage of participants | 1.5 [-15.0 to 18.0] | NA [NA to NA] — NA = Difference in pCR rate between treatments is presented under LCL161 + paclitaxel column (gene expression signature positive) | -2.0 [-12.7 to 8.3] | NA [NA to NA] — NA = Difference in pCR rate between treatments is presented under LCL161 + paclitaxel column (gene expression signature negative)

4. Secondary Outcome: Posterior Distribution of Difference of pCR Rates After Treatment With LCL161 + Paclitaxel Between Patients With Gene Expression Positive and Negative Tumors
Description: To assess whether use of the gene expression signature identifies tumors more likely to respond to treatment with LCL161 and paclitaxel. The measurement type used for this analysis is posterior median and the method of dispersion is Credible Interval (Crl) and not Confidence Interval (CI). 95% Confidence interval is actually 95% credible interval.
Time Frame: 12 weeks
Population: Efficacy Analysis Set 1 (EAS1) are patients who received at least 1 full or partial dose of LCL161 + paclitaxel or of paclitaxel alone with a valid gene expression signature score. Gene expression signature status is derived based on continuous gene expression signature score using cut-off 0.6661(positive: score ≥ 0.6661; negative: score <0.6661)
Measure: Median (95% Confidence Interval); unit: Difference in percentage of participants
Groups:
- LCL161 + Paclitaxel: Patients randomized to the experimental arm who received LCL161 1800 mg once weekly + paclitaxel 80 mg/m2 weekly for 12 weeks.
Arm/Group | LCL161 + Paclitaxel
Number analyzed (Participants) | 105
Difference in percentage of participants | 18.2 [5.0 to 32.4]

5. Secondary Outcome: Posterior Distribution of Difference in pCR Rates After Treatment With Paclitaxel Only Between Gene Expression Positive and Negative Tumors
Description: To assess whether use of the gene expression signature identifies tumors more likely to respond to treatment with paclitaxel only. The measurement type used for this analysis is posterior median and the method of dispersion is Credible Interval (Crl) and not Confidence Interval (CI). 95% Confidence interval is actually 95% credible interval.
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Difference in percentage of participants
Groups:
- Paclitaxel Only: Patients randomized to the control arm who received paclitaxel 80 mg/m2 weekly for 12 weeks.
Arm/Group | Paclitaxel Only
Number analyzed (Participants) | 102
Difference in percentage of participants | 13.3 [-0.4 to 27.5]

6. Secondary Outcome: pCR Rate in Breast After 12 Weeks of Therapy With Single Agent LCL161 and LCL161 + Paclitaxel, Regardless of Gene Signature Status
Description: To assess whether adding LCL161 to weekly paclitaxel enhances the efficacy of paclitaxel in women with triple negative breast cancer regardless of tumor gene expression signature status. This comparison is between the 2 study treatments, regardless of gene signature status. The measurement type used for this analysis is posterior median and the method of dispersion is Credible Interval (Crl) and not Confidence Interval (CI). 95% Confidence interval is actually 95% credible interval.
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Percentage of participants
Groups:
- LCL161 + Paclitaxel: Patients randomized to the experimental arm received LCL161 1800 mg once weekly + paclitaxel 80 mg/m2 weekly for 12 weeks.
Arm/Group | LCL161 + Paclitaxel | Paclitaxel Only
Number analyzed (Participants) | 105 | 102
Percentage of participants | 15.5 [9.6 to 22.8] | 15.7 [9.8 to 23.3]

7. Secondary Outcome: pCR Rate in Breast, Regional Nodes and Axilla
Description: To assess other indicators of disease response for the LCL161 + paclitaxel combination compared to paclitaxel alone. The pCR in breast, regional nodes, and axilla were determined based on the America Joint Committee on Cancer Staging [AJCC] stages T1c, T2, N0-N2, M0) were (AJCC) pathologic staging recorded on the eCRF: a patient was considered to be a responder in breast, regional nodes, and axilla if the pathological complete response was reported for breast and if the regional lymph nodes staging was pN0 (including i-, mol-, mol+).The measurement type used for this analysis is posterior median and the method of dispersion is Credible Interval (Crl) and not Confidence Interval (CI). 95% Confidence interval is actually 95% credible interval.
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LCL161 + Paclitaxel (Gene Expression Signature Positive) | Paclitaxel Only (Gene Expression Signature Positive) | LCL161 + Paclitaxel (Gene Expression Signature Negative) | Paclitaxel Only (Gene Expression Signature Negative)
Number analyzed (Participants) | 50 | 51 | 55 | 51
Percentage of participants | 21.5 [11.8 to 34.0] | 19.1 [10.0 to 31.2] | 6.9 [2.2 to 15.5] | 5.5 [1.4 to 13.9]

8. Secondary Outcome: Rates of Breast Conserving Surgery and Mastectomy - Assessed by Percentage of Patients Who Underwent Breast Conserving Surgery, Masectomy and no Surgery
Description: To assess other indicators of disease response for the LCL161 + paclitaxel combination compared to paclitaxel alone. Rates of breast conserving surgery and mastectomy also contributed to the overall assessment of disease response and were summarized by treatment arm within each gene expression signature status. For this analysis, patients with multicentric breast cancer were excluded, as all patients in this group were expected to be treated with mastectomy.
Time Frame: 16 weeks
Population: EAS1 - patients receiving at least 1 full or partial dose of LCL161 + paclitaxel or of paclitaxel alone with a valid gene expression signature (GES) score. GES status is derived based on continuous GES score using cut-off 0.6661(pos: score ≥ 0.6661; neg: score <0.6661). Patients with multicentric breast cancer were excluded.
Measure: Number; unit: Percentage of participants
Arm/Group | LCL161 + Paclitaxel (Gene Expression Signature Positive) | Paclitaxel Only (Gene Expression Signature Positive) | LCL161 + Paclitaxel (Gene Expression Signature Negative) | Paclitaxel Only (Gene Expression Signature Negative)
Number analyzed (Participants) | 48 | 45 | 51 | 47
Percentage of participants
  Breast Conserving Surgery | 60.4 | 60.0 | 49.0 | 44.7
  Mastectomy | 25.0 | 26.7 | 23.5 | 29.8
  No Surgery | 14.6 | 13.3 | 27.5 | 25.5

9. Secondary Outcome: Caspase 3 Activation in Tumor by Immunohistochemistry (IHC) - EAS1
Description: To evaluate whether combination treatment with LCL161 and paclitaxel is associated with increased apoptosis compared to weekly paclitaxel alone. To evaluate whether combination treatment with LCL161 and paclitaxel was associated with increased apoptosis compared to weekly paclitaxel alone, cleaved caspase 3 activation in tumor by IHC was examined.
  Gene expression signature status is derived based on continuous gene expression signature score using cut-off 0.6661 (positive: score ≥ 0.6661; negative: score <0.6661); cycle = 28 days; each patient had either C1D2 or C1D9
Time Frame: Baseline, Post-baeline at Cycle 1, Day 2 (C1D2) or Cycle 1, Day 9 (C1D9)
Population: Efficacy Analysis Set 1 (EAS1) is patients (pts) who received at least 1 full or partial dose of LCL161 + paclitaxel or of paclitaxel alone with valid gene expression signature score. All pts were considered for analysis (N). Only pts (n) with baseline & post baseline values for the given time point were analyzed for that time point.
Measure: Mean (Standard Deviation); unit: % of positive tumor cells
Arm/Group | LCL161 + Paclitaxel (Gene Expression Signature Positive) | Paclitaxel Only (Gene Expression Signature Positive) | LCL161 + Paclitaxel (Gene Expression Signature Negative) | Paclitaxel Only (Gene Expression Signature Negative)
Number analyzed (Participants) | 50 | 51 | 55 | 51
% of positive tumor cells
  EAS1-Baseline (n: 20, 16, 21, 22) | 1.5 (1.6) | 1.4 (1.3) | 1.4 (3.3) | 2.1 (2.8)
  EAS1 Post-Baseline (n: 20, 16, 21, 22) | 2.6 (1.4) | 2.4 (1.7) | 3.1 (3.1) | 3.1 (6.1)

10. Secondary Outcome: Caspase 3 Activation in Tumor by Immunohistochemistry (IHC) - EAS2
Description: To evaluate whether combination treatment with LCL161 and paclitaxel is associated with increased apoptosis compared to weekly paclitaxel alone. To evaluate whether combination treatment with LCL161 and paclitaxel was associated with increased apoptosis compared to weekly paclitaxel alone, cleaved caspase 3 activation in tumor by IHC was examined. Cycle = 28 days; each patient had either C1D2 or C1D9
Time Frame: Baseline, Post-baeline at Cycle 1, Day 2 or Cycle 1, Day 9
Population: The Efficacy Analysis Set 2 (EAS2) was the same as EAS1 except that the threshold for classifying a patient into the positive gene group was 0.7716. All the EAS2 set participants were considered for the analysis (N). Only participants (n) who had baseline and post baseline values for the given time point were analyzed for that time point.
Measure: Mean (Standard Deviation); unit: % of positive tumor cells
Arm/Group | LCL161 + Paclitaxel (Gene Expression Signature Positive) | Paclitaxel Only (Gene Expression Signature Positive) | LCL161 + Paclitaxel (Gene Expression Signature Negative) | Paclitaxel Only (Gene Expression Signature Negative)
Number analyzed (Participants) | 34 | 29 | 71 | 73
% of positive tumor cells
  EAS2-Baseline (n: 13, 11, 28, 27) | 1.3 (1.8) | 1.6 (1.4) | 1.5 (2.9) | 1.9 (2.6)
  EAS2 Post-Baseline (n:13, 11, 28, 27) | 2.3 (1.4) | 2.7 (1.9) | 3.2 (2.7) | 2.9 (5.6)

11. Secondary Outcome: Pharmacokinetics (PK) Parameters of LCL161 Only for Cmax
Description: To evaluate the PK of LCL161 when given in combination with paclitaxel.
Time Frame: cycle 1 day 1, cycle 4 day 15
Population: The pharmacokinetic analysis set (PAS) consisted of all patients who had at least one blood sample providing evaluable PK data for LCL161. Only sparse/limited PK samples were collected and analyzed.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | LCL161 + Paclitaxel (Gene Expression Signature Negative)
Number analyzed (Participants) | 97
ng/mL
  Cycle 1 Day 1 (n:97) | 2230.00 (1113.41) [186.0 to 4740.0]
  Cycle 4 Day 15 (n:47) | 2310.00 (1161.75) [491.0 to 5250.0]

12. Secondary Outcome: Pharmacokinetics (PK) Parameters of LCL161 Only for Tmax
Description: To evaluate the PK of LCL161 when given in combination with paclitaxel. The pharmacokinetic analysis set (PAS) consisted of all patients who had at least one blood sample providing evaluable PK data for LCL161.
Time Frame: cycle 1 day 1, cycle 4 day 15
Population: as for outcome 11
Measure: Median (Full Range); unit: h
Groups:
- LCL161: Patients randomized to the LCL161 1800 mg once weekly for 12 weeks.
Arm/Group | LCL161
Number analyzed (Participants) | 97
h
  Cycle 1 Day 1 (n:97) | 3.72 (1113.41) [0.5 to 5.8]
  Cycle 4 Day 15 (n:47) | 3.50 (1161.75) [1.0 to 4.2]

13. Secondary Outcome: Pharmacokinetics (PK) Parameters of LCL161 Only for AUClast
Description: To evaluate the PK of LCL161 when given in combination with paclitaxel
Time Frame: cycle 1 day 1, cycle 4 day 15
Population: as for outcome 11
Measure: Median (Full Range); unit: ng*hr/mL
Arm/Group | LCL161
Number analyzed (Participants) | 97
ng*hr/mL
  Cycle 1 Day 1 (n:97) | 5250.70 (1113.41) [465.8 to 13379.0]
  Cycle 4 Day 15 (n:47) | 5522.58 (1161.75) [1070.8 to 13745.5]

ADVERSE EVENTS:
Groups:
- LCL161+PACLITAXEL: Patients randomized to the experimental arm for gene expression signature positive/negative received LCL161 1800 mg once weekly + paclitaxel 80 mg/m2 weekly for 12 weeks. Equal numbers of patients with gene expression signature positive and negative disease were included in each treatment arm.
- PACLITAXEL: Patients randomized to the control arm for gene expression signature positive/negative received paclitaxel 80 mg/m2 weekly for 12 weeks. Equal numbers of patients with gene expression signature positive and negative disease were included in each treatment arm.
Arm/Group | LCL161+PACLITAXEL | PACLITAXEL
Serious Adverse Events (participants affected / at risk) | 45/106 | 7/103
Other Adverse Events (participants affected / at risk) | 106/106 | 101/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCL161+PACLITAXEL (N=106) | PACLITAXEL (N=103)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 2 | 0
Feeling cold (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Pyrexia (General disorders) | 19 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 3 | 1
Atypical pneumonia (Infections and infestations) | 3 | 1
Febrile infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 4 | 0
Pneumonia (Infections and infestations) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Immobile (Social circumstances) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCL161+PACLITAXEL (N=106) | PACLITAXEL (N=103)
Anaemia (Blood and lymphatic system disorders) | 27 | 13
Neutropenia (Blood and lymphatic system disorders) | 33 | 9
Vision blurred (Eye disorders) | 7 | 1
Abdominal pain (Gastrointestinal disorders) | 11 | 8
Abdominal pain upper (Gastrointestinal disorders) | 7 | 4
Constipation (Gastrointestinal disorders) | 24 | 24
Diarrhoea (Gastrointestinal disorders) | 76 | 23
Dry mouth (Gastrointestinal disorders) | 10 | 3
Dyspepsia (Gastrointestinal disorders) | 12 | 10
Nausea (Gastrointestinal disorders) | 45 | 32
Stomatitis (Gastrointestinal disorders) | 26 | 18
Vomiting (Gastrointestinal disorders) | 21 | 16
Asthenia (General disorders) | 16 | 11
Chills (General disorders) | 12 | 4
Fatigue (General disorders) | 48 | 38
Influenza like illness (General disorders) | 6 | 0
Oedema peripheral (General disorders) | 12 | 3
Pyrexia (General disorders) | 44 | 9
Drug hypersensitivity (Immune system disorders) | 8 | 1
Hypersensitivity (Immune system disorders) | 7 | 6
Urinary tract infection (Infections and infestations) | 10 | 3
Procedural pain (Injury, poisoning and procedural complications) | 7 | 9
Alanine aminotransferase increased (Investigations) | 15 | 11
Aspartate aminotransferase increased (Investigations) | 13 | 8
Haemoglobin decreased (Investigations) | 8 | 3
Neutrophil count decreased (Investigations) | 10 | 2
White blood cell count decreased (Investigations) | 8 | 3
Decreased appetite (Metabolism and nutrition disorders) | 12 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 23 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 6
Dizziness (Nervous system disorders) | 12 | 7
Dysgeusia (Nervous system disorders) | 24 | 9
Headache (Nervous system disorders) | 35 | 18
Hypoaesthesia (Nervous system disorders) | 2 | 6
Neuropathy peripheral (Nervous system disorders) | 13 | 28
Neurotoxicity (Nervous system disorders) | 11 | 10
Paraesthesia (Nervous system disorders) | 9 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 25 | 17
Anxiety (Psychiatric disorders) | 8 | 8
Insomnia (Psychiatric disorders) | 22 | 17
Breast pain (Reproductive system and breast disorders) | 9 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 72 | 69
Erythema (Skin and subcutaneous tissue disorders) | 10 | 8
Nail disorder (Skin and subcutaneous tissue disorders) | 5 | 6
Palmar-Plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 28 | 9
Rash (Skin and subcutaneous tissue disorders) | 44 | 27
Flushing (Vascular disorders) | 6 | 7
Hot flush (Vascular disorders) | 17 | 15
Hypertension (Vascular disorders) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.